CLINICAL TRIAL: NCT01749956
Title: A Phase II Study of 5-Fluorouracil (5-FU), Aflibercept, and Radiation for the Preoperative and Adjuvant Treatment of Patients With Stage II/III Rectal Cancer
Brief Title: 5-FU, Aflibercept, and Radiation (RT) for Preoperative and Postoperative Patients With Stage II/III Rectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SCRI Development Innovations, LLC (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCRI GI 168
Record Dates: First submitted 2012-12-12; First posted 2012-12-17 (Estimated); Results first posted 2017-02-07 (Estimated); Last update posted 2017-02-07 (Estimated); Status verified 2016-12

CONDITIONS: Rectal Cancer
Keywords: Rectal Cancer; Chemoradiation; Aflibercept; Surgery
MeSH Terms: conditions — Rectal Neoplasms | interventions — Radiation; aflibercept; Surgical Procedures, Operative; Folfox protocol; Leucovorin; Fluorouracil; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- FOLFOX6/Aflibercept/Radiation/Surgery (Experimental): Preoperative Chemoradiation: (6 weeks)
  * 5-FU: 225 mg/m2 per day by intravenous continuous infusion (IVCI), Days 1 thru 42;
  * Radiation: 50.4 Gy (1.8 Gy/day or 28 fractions) Mon thru Fri, Weeks 1 thru 6;
  * Aflibercept: 4 mg/ kg, via IV infusion, Days 1 and 15.
  Surgery at least 6 weeks after last day of aflibercept: Patients will undergo abdominoperineal or low anterior resection with total mesorectal excision, per standard treatment guidelines.
  Postoperative Chemotherapy and Aflibercept Treatments (four 28-day cycles):
  * Aflibercept (administered first): 4 mg/kg IV for approximately 1 hour (no more than 2 hours) on Days 1 and 15 of each cycle.
  * Modified FOLFOX6:
    * Leucovorin: 400 mg/m2 as a 2-hour infusion prior to 5-FU on Days 1 and 15 of each cycle.
    * Oxaliplatin: 85 mg/m2 IV as a 2-hour infusion prior to 5-FU on Days 1 and 15 of each cycle.
    * 5-FU: 400-mg/m2 bolus for 2 to 4 minutes followed by 2400 mg/m2 for 46 hours on Days 1 and 15 of each cycle.
  Interventions: Radiation: Radiation; Drug: Aflibercept; Procedure: Surgery; Drug: FOLFOX6

INTERVENTIONS:
Radiation: Radiation
Drug: Aflibercept
  Other Names: Eylea; Zaltrap
Procedure: Surgery — Abdominoperineal or low anterior resection with total mesorectal excision, per standard treatment guidelines
Drug: FOLFOX6
  Other Names: Leucovorin (Folinic Acid); 5-Fluorouracil (5-FU; Efudex); Oxaliplatin (Eloxatin)

SUMMARY:
The purpose of this Phase II study will be to investigate the antiangiogenic agent, aflibercept, in combination with chemoradiation as preoperative treatment for patients with stage II/III rectal cancer, followed by 4 months of FOLFOX6 plus aflibercept adjuvantly.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically confirmed stage II or III rectal cancer (adenocarcinoma)
2. Patients must be candidates for preoperative chemoradiation
3. Male or female patients ≥18 years-of-age
4. Eastern Cooperative Oncology Group Performance Status (ECOG PS) score of 0 or 1
5. Adequate hematologic, liver and renal function
6. Male patients willing to use adequate contraceptive measures
7. Female patients who are not of child-bearing potential, and female patients of child-bearing potential who agree to use adequate contraceptive measures, who are not breastfeeding, and who have a negative serum or urine pregnancy test <7 days prior to start of treatment
8. Life expectancy ≥12 weeks
9. Willingness and ability to comply with the trial and follow-up procedures
10. Ability to understand the nature of this trial and give written informed consent.

Exclusion Criteria:

1. Treatment with prior chemotherapy or radiation for rectal cancer.
2. Patients who have received any other investigational agents within the 28 days prior to Day 1 of the study.
3. Known to be human immunodeficiency virus positive or hepatitis B or C positive
4. Women who are pregnant or breastfeeding
5. History of acute myocardial infarction within the previous 6 months, uncontrolled hypertension (blood pressure >150/100 mmHg and/or diastolic blood pressure >100 mmHg), unstable angina, New York Heart Association Grade 2 or greater congestive heart failure, serious cardiac arrhythmia requiring medication (excluding atrial fibrillation), or ≥ Grade 2 peripheral vascular disease.
6. History of hypertensive crisis or hypertensive encephalopathy.
7. History of stroke or transient ischemic attack within the past 6 months.
8. Significant vascular disease (eg, aortic aneurysm requiring surgical repair or recent peripheral arterial thrombosis) within 6 months prior to initiation of therapy.
9. History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within the past 6 months.
10. Patients with symptomatic sensory or peripheral neuropathy (Grade 2 or above).
11. Patients may not have received other agents, either investigational or marketed, that act by primary anti-angiogenic mechanisms.
12. Prior malignancy (except for adequately treated basal-cell or squamous-cell skin cancers, in situ carcinomas, or low grade [Gleason score of 3+3 or less] localized prostate cancer) in the past 5 years.
13. Patients with active concurrent infections or patients with serious underlying medical conditions.
14. Patients receiving full-dose oral or parenteral/SC anticoagulation must be on a stable dosing schedule prior to enrollment; a coumadin dose must be stable for 1 week. If this cannot be achieved, the patient will be ineligible for enrollment.
15. Major surgical procedure or significant traumatic injury within 28 days prior to study initiation, or anticipation of need for major surgical procedure during the course of the study.
16. Core biopsy or other minor surgical procedure, excluding placement of a vascular access device, within 7 days prior to initiation of therapy.
17. Patients with proteinuria, as demonstrated by a urine protein of 2+ or greater at screening. If 2+ or greater proteinuria, a 24-hour urine can be obtained, and if the result is <1 gm/24 hours, the patient is eligible.
18. Any non-healing wound, ulcer, or bone fracture.
19. Any clinical evidence or history of a bleeding diathesis or significant coagulopathy (in the absence of therapeutic anticoagulation).
20. History of hemoptysis (≥½ teaspoon of bright red blood per episode) within 1 month prior to initiation of therapy.
21. History of any other disease, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates use of an investigational drug or that might affect interpretation of the

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2013-01; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johanna C Bendell, M.D., Study Chair — SCRI Development Innovations, LLC
Locations (11):
- United States (11):
  - Florida Cancer Specialists, Fort Myers, Florida
  - Woodlands Medical Specialists, Pensacola, Florida
  - Florida Cancer Specialists, St. Petersburg, Florida
  - Space Coast Cancer Center, Titusville, Florida
  - Baptist Hospital East, Louisville, Kentucky
  - Oncology Hematology Care, Inc., Cincinnati, Ohio
  - Oklahoma University, Oklahoma City, Oklahoma
  - South Carolina Oncology Associates, Columbia, South Carolina
  - Tennessee Oncology - Chattanooga, Chattanooga, Tennessee
  - Tennessee Oncology, PLLC, Nashville, Tennessee
  - Virginia Cancer Institute, Richmond, Virginia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between January 2013 and July 2014, 39 patients with stage II or stage III rectal cancer were enrolled in the trial from multiple sites in the U.S.
Groups:
- FOLFOX6/Aflibercept/Radation/Surgery: Preoperative Chemoradiation (6 weeks): 5-FU: 225 mg/m2 per day by intravenous continuous infusion (IV), Days 1-42; Radiation: 50.4 Gy (1.8 Gy/day) Mon-Fri, Weeks 1 thru 6; Aflibercept: 4 mg/ kg, via IV infusion, Days 1 and 15.
  Surgery (6 weeks from last dose of aflibercep): abdominoperineal or low anterior resection with total mesorectal excision, per standard treatment guidelines.
  Postoperative Chemotherapy and Aflibercept: Aflibercept (administered first): 4 mg/kg IV for approximately 1 hour; Days 1 and 15 of each 28-day cycle; Modified FOLFOX6: Leucovorin: 400 mg/m2 as a 2-hour infusion prior to 5-FU on Days 1 and 15 of each cycle; Oxaliplatin: 85 mg/m2 IV as a 2-hour infusion prior to 5-FU on Days 1 and 15 of each cycle; 5-FU: 400-mg/m2 bolus for 2 to 4 minutes followed by 2400 mg/m2 for 46 hours on Days 1 and 15 of each cycle.
Period: Overall Study
Arm/Group | FOLFOX6/Aflibercept/Radation/Surgery
Started | 39
Completed | 24
Not Completed | 15

BASELINE CHARACTERISTICS:
Population: All enrolled patients
Groups:
- FOLFOX6/Aflibercept/Radation/Surgery: Preoperative Chemoradiation (6 weeks) Surgery (6 weeks from last dose of aflibercept) Postoperative Chemotherapy and aflibercept (four 28-day cycles)
Arm/Group | FOLFOX6/Aflibercept/Radation/Surgery
Number analyzed (Participants) | 39
Age, Continuous [Median (Full Range); unit: years] | 60 [36 to 89]
Gender [Count of Participants; unit: Participants]
  Female | 14
  Male | 25
Race/Ethnicity, Customized [Number; unit: participants]
  White/Caucasian | 38
  Black/African American | 1
Region of Enrollment [Number; unit: participants]
  United States | 39
Carcinoma Stage at Initial Diagnosis [Number; unit: participants] — Eligible patients with a histologically confirmed diagnosis of Stage II or Stage III rectal cancer, staged according to the American Joint Committee on Cancer (AJCC) Staging Manual - Edition 7.
  participants
    Stage II | 12
    Stage III | 27
Baseline ECOG Performance Status [Number; unit: participants] — Eastern Cooperative Oncology Group (ECOG) Performance Status
  0=Fully active, able to carry on all pre-disease performance without restriction
  1. Restricted in physically strenuous activity. Ambulatory and able to carry out work of a light or sedentary nature
  2. Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours
  3. Capable of only limited selfcare; confined to bed or chair more than 50% of waking hours
  4. Completely disabled; cannot carry on any selfcare; totally confined to bed or chair
  5. Dead
  participants
    ECOG Performance Status = 0 | 32
    ECOG Performance Status = 1 | 7
Histologic Grade at Baseline [Number; unit: participants]
  Well differentiated | 4
  Moderately differentiated | 28
  Poorly differentiated | 2
  Could not be assessed | 5

OUTCOME MEASURES:

1. Primary Outcome: Pathologic Complete Response Rate
Description: The Pathologic Complete Response (pCR) Rate is defined as the number of pathologic complete responders among all patients evaluable for response, including evaluable patients who did not proceed to surgery. A pCR is defined as the absence of any residual abnormality detected in a pathological specimen.
Time Frame: Between days 57 and 98 after preoperative chemotherapy
Population: All patients enrolled in the trial who were evaluable for pathologic response. Four patients were not evaluable for response.
Measure: Number; unit: participants
Groups:
- FOLFOX6/Aflibercept/Radiation/Surgery: Preoperative Chemoradiation (6 weeks) Surgery (6 weeks from last dose of aflibercept) Postoperative Chemotherapy and aflibercept (four 28-day cycles)
Arm/Group | FOLFOX6/Aflibercept/Radiation/Surgery
Number analyzed (Participants) | 35
participants | 7

2. Secondary Outcome: Overall Survival
Description: Measured from date of first protocol treatment until date of death.
Time Frame: Every 3 months (±1 month) following documented progression, up to 5 years or death, whichever comes first.
Measure: Median (95% Confidence Interval); unit: participants
Arm/Group | FOLFOX6/Aflibercept/Radiation/Surgery
Number analyzed (Participants) | 39
participants | NA [NA to NA] — Median OS was not reached by time of data analysis.

3. Secondary Outcome: Overall Survival Probability at 6 and 12 Months
Description: The probability of overall survival at 6 months and 12 months from date of first protocol treatment until date of death.
Time Frame: up to 1 year
Measure: Number (95% Confidence Interval); unit: probability
Arm/Group | FOLFOX6/Aflibercept/Radiation/Surgery
Number analyzed (Participants) | 39
probability
  6-month OS probability | 0.97 [0.82 to 0.99]
  12 month OS probability | 0.94 [0.79 to 0.99]

4. Secondary Outcome: Sphincter Preservation Rate
Description: The percentage of patients who had Low Anterior Resection during surgery..
Time Frame: Between days 57 and 98 after preoperative chemotherapy.
Measure: Number; unit: percentage of patients
Arm/Group | FOLFOX6/Aflibercept/Radation/Surgery
Number analyzed (Participants) | 39
percentage of patients | 62

5. Secondary Outcome: Disease-Free Survival
Time Frame: Patients without evidence of progression will be followed every 3 months (±1 month) from date of last dose of study drug during Years 1-2, every 6 months during Years 3-4, and annually thereafter or until disease progression, estimated 5 years.
Population: All evaluable patients.
Measure: Median (95% Confidence Interval); unit: percentage of participants
Arm/Group | FOLFOX6/Aflibercept/Radation/Surgery
Number analyzed (Participants) | 33
percentage of participants | NA [NA to NA] — At a median follow-up of 12 months, median DFS was not reached.

6. Secondary Outcome: Disease Free Survival Probability at 6 and 12 Months
Description: The probability of disease free survival at 6 and 12 months after initiating protocol treatment.
Time Frame: Up to 1 year
Measure: Number (95% Confidence Interval); unit: probability
Arm/Group | FOLFOX6/Aflibercept/Radiation/Surgery
Number analyzed (Participants) | 33
probability
  6-month DFS probability | 0.95 [0.71 to 0.99]
  12-month DFS probability | 0.87 [0.54 to 0.97]

7. Secondary Outcome: The Number of Participants Who Experienced Serious or Non-Serious Adverse Events as a Measure of Safety.
Description: Adverse events and serious adverse events (AEs and SAEs) were graded according to National Cancer Institute Common Technology Criteria for Adverse Events (NCI CTCAE) v4.0. Specific AE and SAE terms are provided in the Adverse Event module.
Time Frame: weekly for 6 weeks pre-op then every 2 weeks post-op, approximately 36 weeks
Population: All patients who received at least one dose of protocol treatment.
Measure: Number; unit: participants
Arm/Group | FOLFOX6/Aflibercept/Radiation/Surgery
Number analyzed (Participants) | 39
participants
  AEs | 38
  SAEs | 9

ADVERSE EVENTS:
Time Frame: From Day 1 of treatment thru 30 days after discontinuation or completion of study treatment, an average of 6 months.
Description: All patients who received at least one dose of protocol treatment during the trial.
Groups:
- FOLFOX6/Aflibercept/Radiation/Surgery: Preoperative Chemoradiation: 5-FU: 225 mg/m2 per day by intravenous continuous infusion (IVCI), Days 1 thru 42; Radiation: 50.4 Gy (1.8 Gy/day or 28 fractions) Mon thru Fri, Weeks 1 thru 6; Aflibercept: 4 mg/ kg, via IV infusion, Days 1 and 15.
  Surgery: Patients will undergo abdominoperineal or low anterior resection with total mesorectal excision, per standard treatment guidelines.
  Postoperative Chemotherapy and Aflibercept Treatments:
  Aflibercept (administered first): 4 mg/kg IV for approximately 1 hour (no more than 2 hours) on Days 1 and 15 of each cycle.
  Modified FOLFOX6:
  * Leucovorin: 400 mg/m2 as a 2-hour infusion prior to 5-FU on Days 1 and 15 of each cycle.
  * Oxaliplatin: 85 mg/m2 IV as a 2-hour infusion prior to 5-FU on Days 1 and 15 of each cycle.
  * 5-FU: 400-mg/m2 bolus for 2 to 4 minutes followed by 2400 mg/m2 for 46 hours on Days 1 and 15 of each cycle.
  Radiation
  Aflibercept
  Surgery: Abdominoperineal or low anterior resectio
Arm/Group | FOLFOX6/Aflibercept/Radiation/Surgery
Serious Adverse Events (participants affected / at risk) | 9/39
Other Adverse Events (participants affected / at risk) | 38/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FOLFOX6/Aflibercept/Radiation/Surgery (N=39)
Pelvic Abscess (Infections and infestations) | 2 (2)
Small Intestinal Obstruction (Gastrointestinal disorders) | 2 (2)
Abscess (Infections and infestations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Device Related Infection (Infections and infestations) | 1 (1)
Embolism Venous (Vascular disorders) | 1 (1)
Enteritis (Gastrointestinal disorders) | 1 (1)
Faecaloma (Gastrointestinal disorders) | 1 (1)
Gastrointestinal Fistula (Gastrointestinal disorders) | 1 (1)
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 (1)
Mucosal Inflammation (General disorders) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (1)
Rectal Ulcer (Gastrointestinal disorders) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | FOLFOX6/Aflibercept/Radiation/Surgery (N=39)
Diarrheoea (Gastrointestinal disorders) | 29
Fatigue (General disorders) | 29
Nausea (Gastrointestinal disorders) | 20
Hypertension (Vascular disorders) | 16
Muscousal Inflammation (General disorders) | 16
Proteinuria (Renal and urinary disorders) | 15
Constipation (Gastrointestinal disorders) | 14
Headache (Nervous system disorders) | 13
Proctalgia (Gastrointestinal disorders) | 12
Anaemia (Blood and lymphatic system disorders) | 11
Decreased Appetite (Metabolism and nutrition disorders) | 10
Dehydration (Metabolism and nutrition disorders) | 9
Neutropenia (Blood and lymphatic system disorders) | 10
Abdominal Pain (Gastrointestinal disorders) | 8
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 8
Thrombocytopenia (Blood and lymphatic system disorders) | 8
Weight Decreased (Investigations) | 8
Dysgeusia (Nervous system disorders) | 7
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 7
Stomatitis (Gastrointestinal disorders) | 7
Vomiting (Gastrointestinal disorders) | 7
Arthralgia (Musculoskeletal and connective tissue disorders) | 6
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 6
Palmar-Plantar Erythrodysaesthesia Syndrome (Skin and subcutaneous tissue disorders) | 6
Rectal Haemorrhage (Gastrointestinal disorders) | 6
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 6
Haematuria (Renal and urinary disorders) | 5
Rash (Skin and subcutaneous tissue disorders) | 5
Temperature Intolerance (General disorders) | 5
Device Related Infection (Infections and infestations) | 5
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4
Hypokalaemia (Metabolism and nutrition disorders) | 4
Leukopenia (Blood and lymphatic system disorders) | 4
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 4
Peripheral Sensory Neuropathy (Nervous system disorders) | 4
Radiation Skin Injury (Injury, poisoning and procedural complications) | 4
Upper Respiratory Tract Infection (Infections and infestations) | 4
Asthenia (General disorders) | 3
Back Pain (Musculoskeletal and connective tissue disorders) | 3
Catheter Site Pain (General disorders) | 3
Dry Skin (Skin and subcutaneous tissue disorders) | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 3
Neutrophil Count Decreased (Investigations) | 3
Paraesthesia (Nervous system disorders) | 3
Dyspepsia (Gastrointestinal disorders) | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 2
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 2
Oral Pain (Gastrointestinal disorders) | 2
Peripheral Neuropathy (Nervous system disorders) | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can review/embargo results communications prior to public release for a period that is >60 days but ≤180 days from date submitted to sponsor, who may require changes to the communication in order to remove specifically identified confidential information (other than study data) and/or delay the proposed publication to enable the sponsor to seek patent protection for inventions. The PI may not publish its results until 18 mos. after the trial has been completed at all sites.